CLINICAL TRIAL: NCT05426291
Title: Is It Possible to Predict Acute Kidney Damage in Patients Undergoing Open Heart Surgery in the Preoperative Period?
Brief Title: Acute Kidney Damage in Patients Undergoing Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Yücel,MD, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: SadiKonuk
Record Dates: First submitted 2022-04-18; First posted 2022-06-21 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Kidney Injury, Acute
Keywords: Open Heart Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — cystatin c level will be checked in the blood sample taken from the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: At least two of the preoperative biomarkers (Mg<0.85 mmol/L, Hgb<8.5 mmol/L, proBNP>480 pg/mL, CRP>5 mg/L) that are thought to be closely related to acute kidney injury after cardiac surgery Group I,
  Interventions: Other: BIOMARKER LEVELS IS IT POSSIBLE TO PREDICT ACUTE RENAL DAMAGE IN THE PREOP PERIOD?
- Group II: Patients who meet at least two of the preoperative biomarkers (Mg>0.85 mmol/L, Hgb>8.5 mmol/L, proBNP<480 pg/mL, CRP<5 mg/L) Group II .
  Interventions: Other: BIOMARKER LEVELS IS IT POSSIBLE TO PREDICT ACUTE RENAL DAMAGE IN THE PREOP PERIOD?

INTERVENTIONS:
Other: BIOMARKER LEVELS IS IT POSSIBLE TO PREDICT ACUTE RENAL DAMAGE IN THE PREOP PERIOD? — In open heart surgery, it will be followed whether acute kidney injury will develop by looking at the biomarkers in the preoperative period.

SUMMARY:
Aimed to determine whether preoperative biomarkers (Mg, Hgb, CRP, ProBNP) would be helpful in the early diagnosis of CSA-AKI (cardiac surgery-related acute kidney injury) in patients undergoing open heart surgery.

DETAILED DESCRIPTION:
An adult patient (aged ≥40 years) with ASA II-IV who was scheduled for elective open heart surgery under cardiopulmonary bypass (CPB) in our clinic between March 1, 2022 and October 30, 2022 will be prospectively included in this study. Patients included in the study will be divided into two groups. At least two of the preoperative biomarkers (Mg<0.85 mmol/L, Hgb<8.5 mmol/L, proBNP>480 pg/mL, CRP>5 mg/L) that are thought to be closely related to acute kidney injury after cardiac surgery Group I, patients who meet at least two of the preoperative biomarkers (Mg>0.85 mmol/L, Hgb>8.5 mmol/L, proBNP<480 pg/mL, CRP<5 mg/L) Group II will be included in the study.Standard monitoring such as electrocardiogram, non-invasive blood pressure and pulsoximetric saturation (SpO2), cerebral oximetry (bSO2, NIRS) will be performed in all open heart surgery patients. To prevent possible kidney damage, colloid fluids and mannitol will not be used as prime solution and replacement fluid in both groups. As in routine open heart surgery, mean arterial pressure (MAP) will be allowed to vary between 55 and 70 mmHg, the volume deficit will be replaced with erythrocyte suspension and/or crystalloid replacement in the form of 500 ml boluses, keeping the hematocrit above 25%. In case of need for a vasoactive agent, dopamine and/or adrenaline infusion is started in the standard open heart surgery procedure. After the operation, the patients are transferred to the cardiovascular surgery intensive care unit (ICU) under the effect of orotracheal intubation and conscious anesthesia. Demographic characteristics of patients (age, gender, height, weight, body mass index, diabetes mellitus, hypertension, peripheral vascular disease, smoking history, hyperlipidemia, atrial fibrillation history, left ventricular ejection fraction) European Cardiac Operative Risk Assessment System (EuroSCORE), baseline bSo2, preoperative magnesium, proBNP, CRP, hemoglobin, serum urea, creatinine value and calculated glomerular filtration rate, cystatin C value, diagnosis, surgical procedure, cardiopulmonary bypass time and cross clamp time will be recorded. Patients with high preoperative Cystatin C levels will be excluded from the study.Serum urea, creatinine concentration and GFR values will be evaluated and recorded at admission to the hospital, one day before surgery, admission to the intensive care unit, and in the mornings of the following 7 days. Cystatin C concentration will be evaluated and recorded the day before surgery, on the first postoperative day (24 hours after surgery).Heart apex, mean arterial pressure, Spo2, bSO2, hemoglobin and hematocrit concentration, lactate, hourly urine volume, diuretic requirement, replaced blood and fluid volume, vasoactive agents before induction of anesthesia {1}, directly before skin incision {2}, after sternum detachment {3}, 20 min after aortic cross clamp {4}, 40 min after aortic cross clamp {5}, 20 min after aortic cross clamp removal {6}, 20 min after CPB release {7}, and {8}eight operations will be recorded in time 60 minutes after leaving the CPB. In the postoperative period, daily total balance, diuretic requirement and vasoactive requirement will be recorded 7 days after the operation. Postoperative complications of the patients, length of stay in the intensive care unit, duration of mechanical ventilation, 28-day mortality will be recorded. The incidence of acute kidney injury will be compared between the patients in Group I and Group II according to the criteria of the Global Result of Improvement of Kidney Disease (KDIGO) criteria and postoperative cystatin C levels during the intraoperative and postoperative period.

ELIGIBILITY:
Mininum Age : 40Years Maximum Age: 85 Years Sex: All Gender Base: No Accepts Healthy Volunteers:No

Criteria:

Inclusion Criteria:

* Elective on-pomp coronary artery bypass

Exclusion Criteria:

* Emergency operation,
* Off pump coronary artery bypass
* Revision (repetitive) operation
* Preoperative acute Renal failure
* Preoperative chronic Renal failure
* Preoperative decompansed heart failure
* Valve replacement surgery

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged ≥40 years,<85 years) with ASA II-IV who were scheduled for elective open heart surgery under cardiopulmonary bypass (CPB) will be prospectively included in this study. Patients included in the study will be divided into two groups. At least two of the preoperative biomarkers (Mg<0.85 mmol/L, Hgb<8.5 mmol/L, proBNP>480 pg/mL, CRP>5 mg/L) that are thought to be closely related to acute kidney injury after cardiac surgery Group I, patients who meet at least two of the preoperative biomarkers (Mg>0.85 mmol/L, Hgb>8.5 mmol/L, proBNP<480 pg/mL, CRP<5 mg/L) Group II will be included in the study.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The requirement of continue venovenous hemodiafiltration (CVVHDF) | Immediately after surgery
  After on pump surgery resulting AKI may require CVVHDF(pH<7.21, urine output < 0.5 ml/kg during 6 hours, potassium > 6 mEq/L)
Predict acute renal failure in on-pomp conary artery bypass via preoperative biomarkers | up to postoperative 28th day
  To detect acute kidney injury in the early period in open heart surgery and to take precautions

SECONDARY OUTCOMES:
The requirement of hemodialysis during postoperative 28 days | up to postoperative 28th day
  After discharging AKI will occur any time line of postoperative period ((pH<7.21, urine output < 0.5 ml/kg,potassium >6 mEq/l)

CONTACTS AND LOCATIONS:
Overall Officials: Gülsüm Oya HERGÜNSEL, Ass. Prof., Study Chair — Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Locations (1):
- BakirkoySadiKonuk Training and Searching Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Associations Between Preoperative Biomarkers and Cardiac Surgery-Associated Acute Kidney Injury in Elderly Patients: A Cohort Study — https://pubmed.ncbi.nlm.nih.gov/34153017/
- See also: Postoperative kidney oxygen saturation as a novel marker for acute kidney injury after adult cardiac surgery — http://doi.org/10.1016/j.jtcvs.2018.09.115